CLINICAL TRIAL: NCT05324592
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase I Trial Comparing the Safety, Pharmacokinetics and Efficacy of 9MW0813 and Aflibercept (EYLEA®) After a Single Dose in Patients With Diabetic Macular Edema (DME)
Brief Title: Safety and Efficacy of 9MW0813 in Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW0813-2020-CP101
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Macular Edema
Keywords: aflibercept; biosimilarity; safety; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW0813 (Experimental)
  Interventions: Drug: 9MW0813
- aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: 9MW0813 — The active ingredient of 9MW0813 injection is recombinant human vascular endothelial growth factor receptor-antibody fusion protein.
  One dose(2mg) of the drug will be injected intravitreously.
  Arms: 9MW0813
Drug: Aflibercept — Aflibercept (trade name: Eylea®/EYLEA®) is an anti-VEGF drug developed by Regeneron/Bayer. It is a fusion protein of human VEGFR1 and VEGFR2 extracellular domains and human immunoglobulin Fc segment genes.
  One dose(2mg) of the drug will be injected intravitreously.
  Other Names: Eylea®
  Arms: aflibercept

SUMMARY:
A multicenter, randomized, double-blind, parallel-controlled phase I trial comparing the safety, pharmacokinetics and efficacy of 9MW0813 and aflibercept (EYLEA®) after a single dose in patients with diabetic macular edema (DME).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel controlled Phase I clinical trial.

The primary objective is to compare the safety of a single intravitreal injection (IVT) of 9MW0813 injection and aflibercept intraocular injection solution (EYLEA®) in DME patients.

The secondary objectives are to comparing the pharmacokinetic profile, immunogenicity and efficacy of a single intravitreal injection (IVT) of 9MW0813 injection and aflibercept intraocular injection solution (EYLEA®) in DME patients.

ELIGIBILITY:
Main inclusion criteria：

1. Diagnosed with type 1 or type 2 diabetes with HbA1c ≤ 11.0%;
2. Use ETDRS chart BCVA ≥ 19 letters and ≤ 73 letters (approximately equivalent to Snellen chart equivalent 20/40 to 20/400);
3. Central retinal thickness (CRT) ≥ 300 μm, (using spectral domain optical coherence tomography);
4. BCVA ≥ 24 letters in the non-study eye (approximately 20/320 equivalent on the Snellen chart).

Main exclusion criteria:

1. with proliferative diabetic retinopathy (PDR), excluding inactive, fibrotic PDR;
2. Vitreous hemorrhage within 30 days before the first administration;
3. Structural retinal damage involving the fovea (such as retinal pigment epithelium (RPE) atrophy, retinal fibrosis, laser scarring, dense hard exudates), or the investigator believes that the study eye has other factors that may hinder vision after macular edema subsides increased retinal damage;
4. Existing ophthalmic conditions other than diabetic retinopathy that cause macular edema or vision changes (such as retinal vein occlusion (RVO), choroidal neovascularization, retinal detachment, macular hole, macular retinal traction, epiretinal membrane, etc.) ;
5. There are iris neovascularization;
6. Uncontrolled glaucoma (defined as intraocular pressure ≥ 25mmHg after anti-glaucoma drug treatment) or glaucoma-causing cup/optic disc ratio of the study eye >0.8 or previous glaucoma filtering surgery (such as trabeculae); excision, sclerectomy, etc.);
7. The investigator believes that the cataract may affect the judgment of the examination or test results, or requires surgical treatment during the test;
8. Aphakia (excluding intraocular lens) or posterior capsule defect (except for YAG laser posterior capsulotomy after intraocular lens implantation within 30 days);
9. History of vitrectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | baseline to week 6

SECONDARY OUTCOMES:
Peak Plasma Concentration（Cmax） of 9MW0813 and aflibercept | baseline to week 6
  Pharmacokinetic measure
Area under the plasma concentration versus time curve (AUC) of 9MW0813 and aflibercept | baseline to week 6
  Pharmacokinetic measure
Immunogenicity of IVT injection of 9MW0813 and aflibercept | baseline to week 6
  Anti-drug antibody (ADA) in serum is detected, ADA-positive samples will be subjected to titer analysis and neutralizing antibody (Nab) analysis
Change from Baseline in Best Corrected Visual Acuity (BCVA) | baseline to week 6
  Change from Baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study(ETDRS) letter score

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing tongren hospital affliated to capital medical university, Beijing, Beijing Municipality, China